CLINICAL TRIAL: NCT00369382
Title: A Randomized Open-Label Study To Compare The Safety And Efficacy Of Conversion From A Calcineurin Inhibitor To Sirolimus Vs Continued Use Of A Calcineurin Inhibitor In Heart Transplant Recipients With Mild-Moderate Impaired Renal Function
Brief Title: Study Of The Safety And Efficacy Of Conversion From A CNI To Sirolimus In Renally-Impaired Heart Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0468E7-408; B1741006 (Other: Pfizer)
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Results first posted 2011-05-23 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Graft Rejection; Kidney Failure
Keywords: Heart Transplant; Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Cyclosporine; Tacrolimus; Cyclosporins; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Group 1: Continuation of CNI regimen
  Interventions: Drug: cyclosporine or tacrolimus
- 2 (Experimental): Group 2: (CNI-Free) Conversion to SRL-based regimen
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: cyclosporine or tacrolimus — Cyclosporine and tacrolimus are provided by the sites and dosed to achieve a target trough level determined by the investigator; therefore, form, dosage, and frequency are site and patient specific. Duration should be 52 weeks on-therapy.
  Other Names: Brand names for cyclosporine are Neoral®, Sandimmune®, and Gengraf®; brand names for tacrolimus are Prograf® and Adagraf™.
  Arms: 1
Drug: sirolimus — Oral (1 and 2 mg) tablets, dosing should be once daily to achieve a target trough level of 7- 15 ng/mL. Duration should be 52 weeks on-therapy.
  Other Names: Rapamune®
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine whether converting from calcineurin inhibitor (CNI) therapy to sirolimus therapy will be more effective than continuing calcineurin inhibitor therapy with respect to renal function in cardiac transplant recipients with mild to moderate renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac transplant recipients age 18 years or older receiving cyclosporine or tacrolimus since the time of transplant.
* 12 months after cardiac transplantation but less than 96 months post-transplantation.

Exclusion Criteria:

* Multiple-organ transplant recipients (such as heart-lung, heart-kidney, or heart after kidney transplant recipients).
* Prior or current use of sirolimus or everolimus unless administration was part of a "CNI holiday" lasting no more than 10 days.
* History of acute rejection within the last 3 months, malignancy within the last 5 years (except for adequately treated basal cell or squamous cell carcinoma of the skin), and human immunodeficiency virus (HIV) patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-09; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (7):
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
- Pfizer Investigational Site, Darlinghurst, New South Wales, Australia
- Pfizer Investigational Site, Vienna, Austria
- Canada (3):
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sainte-Foy, Quebec
- New Zealand (2):
  - Pfizer Investigational Site, Epsom, Auckland
  - Pfizer Investigational Site, Auckland, New Zealand
- Spain (7):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, La Coru?a, La Coru?a
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Barcelona
- Pfizer Investigational Site, Bern, Switzerland

REFERENCES:
- [Derived] Zuckermann A, Keogh A, Crespo-Leiro MG, Mancini D, Vilchez FG, Almenar L, Brozena S, Eisen H, Tai SS, Kushwaha S. Randomized controlled trial of sirolimus conversion in cardiac transplant recipients with renal insufficiency. Am J Transplant. 2012 Sep;12(9):2487-97. doi: 10.1111/j.1600-6143.2012.04131.x. Epub 2012 Jul 9. PMID 22776430
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0468E7-408&StudyName=Study%20Of%20The%20Safety%20And%20Efficacy%20Of%20Conversion%20From%20A%20CNI%20To%20Sirolimus%20In%20Renally-Impaired%20Heart%20Transplant%20Recipients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Actual number of participants randomized was 121; however 5 participants randomized in error. They were withdrawn from study as screen failures, not administered study drug. Participants randomized (121) lower than planned (200); more sites added, time period to enroll extended twice up to 2.5 years. Despite this, final enrollment below planned.
Groups:
- Cyclosporine or Tacrolimus: Continuation of Calcineurin inhibitor (CNI) regimen; included cyclosporine (CsA) or tacrolimus (TAC) which were dosed to achieve a target trough level determined by investigator; therefore, form, dosage, and frequency were site and patient specific. CsA therapy could have been switched to TAC therapy and vice versa, as warranted by clinical circumstances.
- Sirolimus (SRL): Conversion from CNI therapy to Sirolimus: Sirolimus initiated with oral tablets administered once daily (1 to 5 milligrams per day) to achieve target trough of 8-15 nanograms per milliliter (ng/mL). Protocol was later amended to allow target troughs of 7-15 ng/mL for duration of study. CNI discontinued within 8 weeks post randomization.
Period: Overall Study
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Started | 59 | 57
Received Treatment | 57 | 57
Completed Assigned Treatment Regimen | 48 | 33
Completed | 49 | 54
Not Completed | 10 | 3
Not completed — Death | 0 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Randomized, not treated | 2 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL) | Total
Number analyzed (Participants) | 59 | 57 | 116
Age Continuous [Mean (Standard Deviation); unit: years] | 58.93 (8.01) | 57.40 (9.42) | 58.18 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 54 | 45 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Calculated Creatinine Clearance (Cockcroft-Gault Equation) at 52 Weeks Post-randomization
Description: Creatinine Clearance (CC) calculated using Cockcroft-Gault equation, adjusted for body surface area. Calculated CC: method to approximate kidney function. It measures rate creatinine (substance formed from metabolism of creatine) is cleared from blood by kidneys. Normal adult creatinine clearance is greater than or equal to (≥) 90 milliliters per minute per 1.73 meters squared (mL/min/1.73m^2). Change from baseline=CC at Week 52 minus CC at baseline where higher scores represented improved renal function; Least squares mean adjusted for baseline calculated creatinine clearance and center.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population: all randomized participants; all available data (on-therapy and off-therapy) included; Last observation carried forward (LOCF) for data missing due to skipped visits or participant withdrawal from study. Number of participants analyzed (N)=those with all measurements required for calculated creatinine clearance.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 59 | 56
mL/min/1.73m^2 | -1.35 (1.18) | 3.03 (1.29)
Statistical Analysis 1: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 52; Test type: Superiority or Other; p = 0.004, ANCOVA — two-sided alpha = 0.05; Analysis of covariance (ANCOVA) with baseline creatinine clearance (Cockcroft-Gault) as a covariate and treatment group and center as factors

2. Primary Outcome: Calculated Creatinine Clearance (Cockcroft-Gault Equation) at Baseline
Description: Creatinine clearance at baseline calculated using Cockcroft-Gault equation and adjusted for body surface area. Calculated CC: method to approximate kidney function. It measures rate creatinine (substance formed from metabolism of creatine) is cleared from blood by kidneys. Normal adult creatinine clearance is ≥ 90 mL/min/1.73m^2.
Time Frame: Baseline
Population: ITT; N=participants with all measurements required for calculated creatinine clearance.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 59 | 56
mL/min/1.73m^2 | 57.09 (11.96) | 57.75 (14.04)

3. Secondary Outcome: Change From Baseline in Calculated Creatinine Clearance (Cockcroft-Gault Equation) at 4, 16, 24, 32, and 40 Weeks Post-randomization
Description: Creatinine Clearance (CC) calculated using Cockcroft-Gault equation, adjusted for body surface area. Calculated CC: method to approximate kidney function. It measures rate creatinine (substance formed from metabolism of creatine) is cleared from blood by kidneys. Normal adult creatinine clearance is ≥ 90 mL/min/1.73m^2. Change from baseline=CC at Week X minus CC at baseline where higher scores represented improved renal function; Least squares mean adjusted for baseline calculated creatinine clearance and center.
Time Frame: Baseline and Weeks 4, 16, 24, 32, and 40
Population: ITT; All available data (on-therapy and off-therapy) were included; LOCF for data points missing due to skipped visits or participant withdrawal from study; N=participants with all measurements required for calculated creatinine clearance.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 59 | 56
mL/min/1.73m^2
  Week 4 | -0.20 (1.06) | 2.96 (1.16)
  Week 16 | -2.16 (1.37) | 3.79 (1.50)
  Week 24 | -1.91 (1.28) | 2.15 (1.40)
  Week 32 | -0.76 (1.32) | 2.22 (1.45)
  Week 40 | 0.34 (1.39) | 2.70 (1.52)
Statistical Analysis 1: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 4; Test type: Superiority or Other; p = 0.018, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (Cockcroft-Gault) as a covariate and treatment group and center as factors
Statistical Analysis 2: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 16; Test type: Superiority or Other; p < .001, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (Cockcroft-Gault) as a covariate and treatment group and center as factors
Statistical Analysis 3: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 24; Test type: Superiority or Other; p = 0.012, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (Cockcroft-Gault) as a covariate and treatment group and center as factors
Statistical Analysis 4: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 32; Test type: Superiority or Other; p = 0.072, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (Cockcroft-Gault) as a covariate and treatment group and center as factors
Statistical Analysis 5: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 40; Test type: Superiority or Other; p = 0.175, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (Cockcroft-Gault) as a covariate and treatment group and center as factors

4. Secondary Outcome: Change From Baseline in Calculated Creatinine Clearance (Modification of Diet in Renal Disease [MDRD] Equation) at 4, 16, 24, 32, 40 and 52 Weeks Post-randomization
Description: Creatinine clearance calculated using MDRD equation. Normal adult creatinine clearance is ≥ 90 mL/min/1.73m^2. Change from baseline=CC at Week X minus CC at baseline where higher scores represented improved renal function. Least squares mean adjusted for baseline calculated creatinine clearance (MDRD) and center.
Time Frame: Baseline and Weeks 4, 16, 24, 32, 40 and 52
Population: ITT; All available data (on-therapy and off-therapy) were included; LOCF for data points missing due to skipped visits or participant withdrawal from study.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 59 | 57
mL/min/1.73m^2
  Week 4 | -0.00 (1.16) | 3.18 (1.25)
  Week 16 | -1.92 (1.40) | 4.30 (1.51)
  Week 24 | -1.47 (1.36) | 2.54 (1.47)
  Week 32 | -0.15 (1.43) | 2.44 (1.54)
  Week 40 | 0.69 (1.52) | 2.69 (1.64)
  Week 52 | -0.90 (1.26) | 3.26 (1.36)
Statistical Analysis 1: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 4; Test type: Superiority or Other; p = 0.031, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (MDRD) as a covariate and treatment group and center as factors
Statistical Analysis 2: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (MDRD) as a covariate and treatment group and center as factors
Statistical Analysis 3: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 24; Test type: Superiority or Other; p = 0.020, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (MDRD) as a covariate and treatment group and center as factors
Statistical Analysis 4: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 32; Test type: Superiority or Other; p = 0.151, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (MDRD) as a covariate and treatment group and center as factors
Statistical Analysis 5: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 40; Test type: Superiority or Other; p = 0.295, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (MDRD) as a covariate and treatment group and center as factors
Statistical Analysis 6: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 52; Test type: Superiority or Other; p = 0.010, ANCOVA — alpha is unadjusted; ANCOVA with baseline creatinine clearance (MDRD) as a covariate and treatment group and center as factors

5. Secondary Outcome: Calculated Creatinine Clearance (Modification of Diet in Renal Disease [MDRD] Equation) at Baseline
Description: Creatinine clearance calculated using MDRD equation. Calculated CC: method to approximate kidney function. It measures rate creatinine (substance formed from metabolism of creatine) is cleared from blood by kidneys. Normal adult creatinine clearance is ≥ 90 mL/min/1.73m^2.
Time Frame: Baseline
Population: ITT.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 59 | 57
mL/min/1.73m^2 | 55.39 (12.84) | 54.47 (14.14)

6. Secondary Outcome: Change From Baseline in Serum Creatinine Level at 4, 16, 24, 32, 40, and 52 Weeks Post-randomization
Description: Serum creatinine is an indicator of kidney function. Creatinine is a substance formed from the metabolism of creatine, commonly found in blood, urine, and muscle tissue. It is removed from the blood by the kidneys and excreted in urine. Normal adult blood levels of creatinine=45 to 90 micromoles per liter (mcmol/L) for females, 60 to 110 mcmol/L for males, however normal values are age-dependent. Change from baseline=creatinine level at Week x minus baseline level where higher scores represented decreased kidney function. Least squares mean adjusted for treatment group and center.
Time Frame: Baseline and Weeks 4, 16, 24, 32, 40, and 52
Population: ITT, All available data (on-therapy and off-therapy) were included; LOCF for data points missing due to skipped visits or participant withdrawal from study.
Measure: Least Squares Mean (Standard Error); unit: mcmol/L
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 59 | 57
mcmol/L
  Week 4 | 1.68 (2.00) | -4.95 (2.15)
  Week 16 | 7.96 (2.62) | -5.52 (2.82)
  Week 24 | 8.02 (2.21) | -0.89 (2.37)
  Week 32 | 4.08 (2.52) | -2.80 (2.71)
  Week 40 | 2.44 (2.70) | 2.81 (2.90)
  Week 52 | 4.76 (2.22) | -4.39 (2.39)
Statistical Analysis 1: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 4; Test type: Superiority or Other; p = 0.009, ANCOVA — alpha is unadjusted; ANCOVA with baseline serum creatinine as a covariate and treatment group and center as factors
Statistical Analysis 2: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA — alpha is unadjusted; ANCOVA with baseline serum creatinine as a covariate and treatment group and center as factors
Statistical Analysis 3: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 24; Test type: Superiority or Other; p = 0.002, ANCOVA — alpha is unadjusted; ANCOVA with baseline serum creatinine as a covariate and treatment group and center as factors
Statistical Analysis 4: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 32; Test type: Superiority or Other; p = 0.030, ANCOVA — alpha is unadjusted; ANCOVA with baseline serum creatinine as a covariate and treatment group and center as factors
Statistical Analysis 5: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 40; Test type: Superiority or Other; p = 0.121, ANCOVA — alpha is unadjusted; ANCOVA with baseline serum creatinine as a covariate and treatment group and center as factors
Statistical Analysis 6: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Change from baseline to Week 52; Test type: Superiority or Other; p = 0.001, ANCOVA — alpha is unadjusted; ANCOVA with baseline serum creatinine as a covariate and treatment group and center as factors

7. Secondary Outcome: Serum Creatinine Level at Baseline
Description: Serum creatinine is an indicator of kidney function. Creatinine is a substance formed from the metabolism of creatine, commonly found in blood, urine, and muscle tissue. It is removed from the blood by the kidneys and excreted in urine.
Time Frame: Baseline
Population: ITT.
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 59 | 57
mcmol/L | 125.42 (23.15) | 126.21 (29.63)

8. Secondary Outcome: Annual Change in Calculated Creatinine Clearance (Cockcroft-Gault Equation)
Description: The change in creatinine clearance over time assessed using the random coefficient slope of the regression line with creatinine clearance as the dependent variable and study day as the independent variable. Time points calculated as study days, relative to time of randomization of study medication. Observed data multiplied by a scale factor of 365 to express an annual change.
Time Frame: Baseline to discontinuation (up to Week 52)
Population: ITT; N=participants with all measurements required for calculated creatinine clearance. All observed data up to the point of discontinuation of the study were used.
Measure: Number (95% Confidence Interval); unit: mL/min/1.73m^2
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 59 | 56
mL/min/1.73m^2 | -0.740 [-2.921 to 1.441] | 1.571 [-0.447 to 3.588]
Statistical Analysis 1: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Test type: Superiority or Other; p = 0.126, Random coefficient model — alpha is unadjusted; slope difference (CNI - SRL) = -2.311, 95% CI 2-sided [-5.282 to 0.660] — Random coefficient model with each participant's creatinine clearance function of time on treatment; intra-subject regression coefficients considered random

9. Secondary Outcome: Overall Survival (OS)
Description: Survival time from the start of study treatment to date of death due to any cause, censored at the last visit if no death. Death was determined from the Death report. The distribution of time to death was to be estimated using Kaplan-Meier method and compared between treatment groups with a proportional hazard model. The number and percent of survival at 6 and 12 months were to be reported.
Time Frame: Baseline until death (up to Week 56)
Population: Safety population: all randomized participants who received at least 1 dose of study medication; not analyzed by Kaplan-Meier because number of events limited to 2 deaths in the sirolimus group.
Measure: Number; unit: Weeks
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Acute Rejection
Description: Based on International Society for Heart and Lung Transplantation [ISHLT] 1990 criteria: rejections Grade 3A or higher, rejection accompanied by hemodynamic compromise or requiring treatment. Grade 3A or higher included: multifocal aggressive infiltrates and/or myocyte damage, diffuse inflammatory process with necrosis, diffuse aggressive polymorphus with necrosis, increased infiltrates, and changes in edema, hemorrhage, or vasculitis. Biopsies performed for clinically suspected rejection (for cause), site's standard of care (site protocol biopsy), or protocol mandated.
Time Frame: Baseline to Week 52
Population: Safety population; n=number of participants analyzed for the specified type of biopsy.
Measure: Number; unit: Participants
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 57 | 57
Participants
  For cause biopsies (n=57, 57) | 1 | 5
  Standard of Care biopsies (n=11, 11) | 0 | 2
  Protocol mandated biopsies (n=0, 39) | NA — Only participants randomized to sirolimus had protocol mandated biopsies 2 to 6 weeks after conversion to sirolimus. | 7
Statistical Analysis 1: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); For-cause Biopsy-Confirmed Acute Rejection compared between treatment groups; Test type: Superiority or Other; p = 0.206, Fisher Exact — alpha is unadjusted
Statistical Analysis 2: Comparison: Cyclosporine or Tacrolimus vs Sirolimus (SRL); Standard of Care Biopsy-Confirmed Acute Rejection compared between treatment groups; Test type: Superiority or Other; p = 0.476, Fisher Exact — alpha is unadjusted

11. Secondary Outcome: Number of Participants With Biopsy-confirmed Acute Rejection by Severity
Description: Severity of acute rejection summarized using revised 2005 ISHLT criteria. Grade 0R: no rejection, Grade 1R: Focal (perivascular or interstitial) infiltrate without necrosis, diffuse but sparse infiltrate without necrosis, or one focus only with aggressive infiltration and/or focal myocyte damage, Grade 2R:Multifocal aggressive infiltrates and/or myocyte damage, and Grade 3R:Diffuse inflammatory process with necrosis, or diffuse aggressive polymorphous with necrosis, increased infiltrate, changes in edema, hemorrhage and vasculitis.
Time Frame: Baseline to Week 52
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 57 | 57
Participants
  Grade 0R protocol mandated | NA — Only participants randomized to the Sirolimus group were required to have protocol mandated biopsies. | 0
  Grade 0R for cause | 0 | 0
  Grade 0R site protocol | 0 | 0
  Grade 1R protocol mandated | NA — Only participants randomized to the Sirolimus group were required to have protocol mandated biopsies. | 0
  Grade 1R for cause | 0 | 0
  Grade 1R site protocol | 0 | 0
  Grade 2R protocol mandated | NA — Only participants randomized to the Sirolimus group were required to have protocol mandated biopsies. | 6
  Grade 2R for cause | 0 | 4
  Grade 2R site protocol | 0 | 1
  Grade 3R protocol mandated | NA — Only participants randomized to the Sirolimus group were required to have protocol mandated biopsies. | 1
  Grade 3R for cause | 1 | 1
  Grade 3R site protocol | 0 | 1

12. Secondary Outcome: Time to First Acute Rejection
Description: Time from baseline to first biopsy-confirmed acute rejection defined as any of the following (based on ISHLT 1990 criteria): all rejections Grade 3A or higher, any rejection accompanied by hemodynamic compromise, or any rejection requiring treatment. ISHLT Grade 3A or higher included: Multifocal aggressive infiltrates and/or myocyte damage, diffuse inflammatory process with necrosis, diffuse aggressive polymorphus with necrosis, increased infiltrates, and changes in edema, hemorrhage, or vasculitis.
Time Frame: Baseline to Week 52
Population: Safety population; not analyzed because actual start date of rejection was unknown for those diagnosed by site protocol (SOC) biopsy and protocol-required biopsy.
Measure: Number; unit: Weeks
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants Requiring Antibody Use in Treatment of Acute Rejection
Description: Number of participants requiring antilymphocyte antibody therapy with suspected or biopsy-proven, steroid-resistant, acute rejection with or without hemodynamic compromise. Acute rejection based on ISHLT 1990 criteria: all rejections Grade 3A or higher, any rejection accompanied by hemodynamic compromise, or any rejection requiring treatment. ISHLT Grade 3A or higher included: Multifocal aggressive infiltrates and/or myocyte damage, diffuse inflammatory process with necrosis, diffuse aggressive polymorphus with necrosis, increased infiltrates, and changes in edema, hemorrhage, or vasculitis.
Time Frame: Baseline to Week 52
Population: Safety population; N=participants who had biopsy-confirmed acute rejection.
Measure: Number; unit: Participants
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Number analyzed (Participants) | 1 | 14
Participants | 1 | 0

14. Secondary Outcome: Number of Participants in Sirolimus Treatment Group Requiring Conversion Back to CNI Therapy
Time Frame: Baseline up to Week 52
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Sirolimus (SRL)
Number analyzed (Participants) | 57
Participants | 21

ADVERSE EVENTS:
Time Frame: Baseline up to Week 56
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Cyclosporine or Tacrolimus | Sirolimus (SRL)
Serious Adverse Events (participants affected / at risk) | 13/57 | 30/57
Other Adverse Events (participants affected / at risk) | 40/57 | 54/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporine or Tacrolimus (N=57) | Sirolimus (SRL) (N=57)
Abdominal pain (General disorders) | 1 | 1 — Body as a Whole
Asthenia (General disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Lab test abnormal (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Transplant rejection (General disorders) | 1 | 13 — Multiple reasons for cardiac biopsies. Refer to outcome measure 10.
Angina pectoris (Cardiac disorders) | 1 | 0 — Cardiovascular System
Arrhythmia (Cardiac disorders) | 0 | 1
Cerebral ischemia (Cardiac disorders) | 0 | 1
Endocarditis (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Syncope (Cardiac disorders) | 1 | 0
Biliary pain (Gastrointestinal disorders) | 0 | 1 — Digestive System
Cholelithiasis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal carcinoma (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Liver function tests abnormal (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 — Hemic and lymphatic system
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 — Musculoskeletal system
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Confusion (Nervous system disorders) | 0 | 1 — Nervous system
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Respiratory system
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 0 — Skin and appendages
Skin carcinoma (Skin and subcutaneous tissue disorders) | 3 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cyclosporine or Tacrolimus (N=57) | Sirolimus (SRL) (N=57)
Abdominal pain (General disorders) | 3 | 7 — Body as a Whole
Accidental injury (General disorders) | 0 | 4
Asthenia (General disorders) | 5 | 5
Back pain (General disorders) | 2 | 4
Chest pain (General disorders) | 0 | 3
Face edema (General disorders) | 1 | 5
Fever (General disorders) | 1 | 4
Generalized edema (General disorders) | 1 | 3
Headache (General disorders) | 2 | 8
Pain (General disorders) | 1 | 5
Transplant rejection (General disorders) | 1 | 4 — Multiple reasons for cardiac biopsies. Refer to outcome measure 10.
Hypertension (Cardiac disorders) | 2 | 7 — Cardiovascular system
Tachycardia sinus (Cardiac disorders) | 1 | 3
Anorexia (Gastrointestinal disorders) | 0 | 3 — Digestive system
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 8
Diarrhea (Gastrointestinal disorders) | 6 | 15
Liver function tests abnormal (Gastrointestinal disorders) | 0 | 3
Mouth ulceration (Gastrointestinal disorders) | 0 | 6
Nausea (Gastrointestinal disorders) | 5 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 3
Anemia (Blood and lymphatic system disorders) | 0 | 5 — Hemic and Lymphatic system
Ecchymosis (Blood and lymphatic system disorders) | 0 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 4
Creatinine increased (Metabolism and nutrition disorders) | 3 | 0 — Metabolic and Nutritional
Gout (Metabolism and nutrition disorders) | 1 | 4
Healing abnormal (Metabolism and nutrition disorders) | 1 | 3
Hypercholesteremia (Metabolism and nutrition disorders) | 1 | 6
Hyperlipemia (Metabolism and nutrition disorders) | 1 | 6
Peripheral edema (Metabolism and nutrition disorders) | 9 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6 — Musculoskeletal system
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Anxiety (Nervous system disorders) | 0 | 3 — Nervous system
Depression (Nervous system disorders) | 0 | 3
Dizziness (Nervous system disorders) | 4 | 5
Insomnia (Nervous system disorders) | 1 | 4
Somnolence (Nervous system disorders) | 1 | 5
Cough increased (Respiratory, thoracic and mediastinal disorders) | 6 | 5 — Respiratory system
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 8 — Skin and Appendages
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 16
Sweating (Skin and subcutaneous tissue disorders) | 1 | 4
Eye pruritus (Eye disorders) | 0 | 3 — Special senses
Uterine fibroids enlarged (Renal and urinary disorders) | 1/5 | 0/12 — Urogenital system
Uterine hemorrhage (Renal and urinary disorders) | 1/5 | 0/12
Infection (General disorders) | 0 | 5 — Body as a whole
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 — Due to infection, Respiratory system
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Herpes simplex (Skin and subcutaneous tissue disorders) | 0 | 4 — Skin and Appendages
Herpes zoster (Skin and subcutaneous tissue disorders) | 4 | 5
Skin carcinoma (Skin and subcutaneous tissue disorders) | 1 | 3 — Skin and Appendages

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.